CLINICAL TRIAL: NCT04914845
Title: A Phase 1 Open-label Study of KPT-9274 in Patients With Relapsed and Refractory Acute Myeloid Leukemia
Brief Title: KPT-9274 in Patients With Relapsed and Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 20-2350.cc; NCI-2021-08786 (Other: CTRP); KPT-9274 (Other: Karyopharm Theraeutics Inc.)
Record Dates: First submitted 2021-05-25; First posted 2021-06-07 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — KPT-9274

STUDY DESIGN:
Intervention Model Description: During dose escalation, patients will receive oral KPT-9274 three times a week every other day (Days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26) during each 28-day cycle, and the first dose cohort will be 30 mg. Subsequent dose escalation cohorts, as well as a de-escalation cohort, will be administered. Dose escalation will continue until the MTD is determined. The MTD is defined as the highest dose at which ≤1 patient experiences a DLT in Cycle 1. A RP2D equal to or less than the MTD will be declared and used for the Dose Expansion Phase, if conducted.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- De-escalation Cohort; 20mg (Active Comparator): For the purposes of dose escalation decisions, a standard 3+3 dose escalation design will be used.The initial cohort, Cohort 1, will consist of 3 enrolled patients who will be treated at 30 mg. If the MTD is exceeded at cohort 1, de-escalation to cohort 0 (20 mg) will occur. If the MTD is not exceeded in cohort 1, dose escalation will continue based on a standard 3+3 design at the dose levels.
  Interventions: Drug: KPT-9274
- Cohort 1; 30 mg (Active Comparator): The initial cohort, Cohort 1, will consist of 3 enrolled patients who will be treated at 30 mg.
  Interventions: Drug: KPT-9274
- Cohort 2; 40mg (Active Comparator): Dose escalation to 40 mg after initial cohort (Cohort 1) after a minimum of 1 cycle of treatment, defined as receiving ≥75% of KPT-9274 doses during Cycle 1 (e.g., ≥9 of 12 doses in the 3 doses/week schedule), or have a DLT within the first cycle of treatment to be evaluable for dose escalation decisions.
  Interventions: Drug: KPT-9274
- Cohort 3; 60mg (Active Comparator): Dose escalation to 60 mg after initial cohort (Cohort 1) after a minimum of 1 cycle of treatment, defined as receiving ≥75% of KPT-9274 doses during Cycle 1 (e.g., ≥9 of 12 doses in the 3 doses/week schedule), or have a DLT within the first cycle of treatment to be evaluable for dose escalation decisions.
  Interventions: Drug: KPT-9274
- Cohort 4; 80mg (Active Comparator): Dose escalation to 80 mg after initial cohort (Cohort 1) after a minimum of 1 cycle of treatment, defined as receiving ≥75% of KPT-9274 doses during Cycle 1 (e.g., ≥9 of 12 doses in the 3 doses/week schedule), or have a DLT within the first cycle of treatment to be evaluable for dose escalation decisions.
  Interventions: Drug: KPT-9274
- Cohort 5; 100mg (Active Comparator): Dose escalation to 100 mg after initial cohort (Cohort 1) after a minimum of 1 cycle of treatment, defined as receiving ≥75% of KPT-9274 doses during Cycle 1 (e.g., ≥9 of 12 doses in the 3 doses/week schedule), or have a DLT within the first cycle of treatment to be evaluable for dose escalation decisions.
  Interventions: Drug: KPT-9274

INTERVENTIONS:
Drug: KPT-9274 — KPT-9274 is a first-in-class orally bioavailable, non-competitive, small molecule, dual modulator of p21 protein (Cdc42/Rac)-activated kinase 4 (PAK4) and nicotinamide phosphoribosyltransferase /PBEF/visfatin (NAMPT). NAMPT is the rate-limiting enzyme in the metabolic scavenging pathway that utilizes nicotinamide to replenish nicotinamide adenine dinucleotide (NAD), an essential metabolic cofactor and second messenger. Recent investigations have shown that in in vitro and in vivo models, NAMPT is uniquely essential for relapsed or refractory AML stem cells. Targeting relapsed AML stem cells, through targeting of NAMPT, may allow for a promising therapeutic opportunity for patients with relapsed or refractory AML.

SUMMARY:
This study will evaluate the safety and tolerability of oral KPT-9274 for the treatment of patients with relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
KPT-9274 is a first-in-class orally bioavailable, non-competitive, small molecule, dual modulator of p21 protein (Cdc42/Rac)-activated kinase 4 (PAK4) and nicotinamide phosphoribosyltransferase /PBEF/visfatin (NAMPT). NAMPT is the rate-limiting enzyme in the metabolic scavenging pathway that utilizes nicotinamide to replenish nicotinamide adenine dinucleotide (NAD), an essential metabolic cofactor and second messenger. Recent investigations have shown that in in vitro and in vivo models, NAMPT is uniquely essential for relapsed or refractory AML stem cells. Targeting relapsed AML stem cells, through targeting of NAMPT, may allow for a promising therapeutic opportunity for patients with relapsed or refractory AML.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study related procedures required solely for this research study.
2. Age ≥18 years.
3. Patients with WHO-confirmed non-APL AML who have not responded to or relapsed after at least one prior therapy and for whom no standard therapy that may provide clinical benefit is available.
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
5. Adequate hepatic function:

   * Total bilirubin < 1.5 times the upper limit of normal (ULN) (except patients with Gilbert's syndrome [hereditary indirect hyperbilirubinemia], subjects with Gilbert's syndrome, total bilirubin needs to be ≤ 4 x ULN).
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN (except patients with known liver involvement of their AML who must have AST and ALT ≤ 5.0 times ULN).
6. Adequate renal function: estimated creatinine clearance of ≥ 60 mL/min, calculated using CKD-EPI Creatinine Equation (2021). https://www.kidney.org/content/ckd-epi-creatinine-equation-2021
7. Female patients of child-bearing potential must agree to use dual methods of contraception (including one highly effective and one effective method of contraception) and have a negative serum pregnancy test at Screening. For both male and female patients, effective methods of contraception must be used throughout the study and for 3 months following the last dose.

   1. Fertile female patients must agree to refrain from egg donation from first dose until at least 3 months following the last dose of KPT-9724.
   2. Women should not breastfeed during treatment with KPT-9724 and for 2 weeks after the last dose.
8. 8. Male patients must use 2 highly effective methods of contraception if sexually active with a female of child-bearing potential, during treatment with KPT-9724, during a period of 2 weeks (5 half-lives) after the last dose of KPT-9724 plus a period of 3 months. (for 3.5 months after their last dose of KPT-9724). Fertile male patients must agree to refrain from sperm donation from first dose until at least 3.5 months following the last dose of KPT-9724.

Exclusion Criteria:

1. Female patients who are pregnant or lactating.
2. Radiation, chemotherapy, immunotherapy or any other anticancer therapy, including investigational anti-cancer therapy ≤ 2 weeks prior to C1D1. Hydroxyurea is not considered an anti-cancer therapy.
3. Patients who have not recovered or stabilized (Grade 1 or to their baseline for non-hematologic toxicities) from toxicities related to their previous treatment, except for alopecia.
4. White blood cell count ≥25x109/L (hydroxyurea or leukapheresis permitted to reduce to below the exclusion criteria threshold and allow eligibility)
5. Patients with known active central nervous system (CNS) disease
6. Clinically significant severe heart disease
7. Subjects with uncontrolled systemic fungal, bacterial, viral or other infection despite appropriate antibiotics or other treatment.
8. Known, active hepatitis A, B, or C infection; or known to be positive for HCV RNA or HBsAg (HBV surface antigen). Testing is not required.
9. Patients with significantly diseased or obstructed gastrointestinal tract or uncontrolled vomiting or diarrhea that could interfere with the absorption of KPT-9274.
10. Serious psychiatric or medical conditions that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pollyea, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jones CL, Stevens BM, Pollyea DA, Culp-Hill R, Reisz JA, Nemkov T, Gehrke S, Gamboni F, Krug A, Winters A, Pei S, Gustafson A, Ye H, Inguva A, Amaya M, Minhajuddin M, Abbott D, Becker MW, DeGregori J, Smith CA, D'Alessandro A, Jordan CT. Nicotinamide Metabolism Mediates Resistance to Venetoclax in Relapsed Acute Myeloid Leukemia Stem Cells. Cell Stem Cell. 2020 Nov 5;27(5):748-764.e4. doi: 10.1016/j.stem.2020.07.021. Epub 2020 Aug 20. PMID 32822582

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | De-escalation Cohort; 20mg | Cohort 1; 30 mg | Cohort 2; 40mg | Cohort 3; 60mg | Cohort 4; 80mg | Cohort 5; 100mg
Started | 0 | 5 | 7 | 4 | 0 | 0
Completed | 0 | 5 | 7 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients de-escalated lower than cohort 1 dose. Due to DLTs, no patients treated at cohort 4 or 5 dose level.
Groups:
- Total: Total of all reporting groups
Arm/Group | De-escalation Cohort; 20mg | Cohort 1; 30 mg | Cohort 2; 40mg | Cohort 3; 60mg | Cohort 4; 80mg | Cohort 5; 100mg | Total
Number analyzed (Participants) | 0 | 5 | 7 | 4 | 0 | 0 | 16
Age, Customized [Count of Participants; unit: Participants]
  Under 18 years of age | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 years of age or older | 0 | 5 | 7 | 4 | 0 | 0 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 3 | 1 |  |  | 4
  Male |  | 5 | 4 | 3 |  |  | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Dose escalation will continue until the MTD is determined. The MTD is defined as the highest dose at which ≤1 patient experiences a DLT in Cycle 1. Count of participants who did not experience a DLT are listed in outcome measure data table.
Time Frame: 28 days
Population: No descalation cohort less than cohort 1 dose was needed. Due to DLTs, no patients enrolled to cohort 4 or 5.
Measure: Number; unit: participants
Arm/Group | De-escalation Cohort; 20mg | Cohort 1; 30 mg | Cohort 2; 40mg | Cohort 3; 60mg | Cohort 4; 80mg | Cohort 5; 100mg
Number analyzed (Participants) | 0 | 5 | 7 | 4 | 0 | 0
participants |  | 5 | 5 | 2 |  |
Statistical Analysis 1: Comparison: De-escalation Cohort; 20mg vs Cohort 1; 30 mg vs Cohort 2; 40mg vs Cohort 3; 60mg vs Cohort 4; 80mg vs Cohort 5; 100mg; MTD was determined to be 30 mg; Test type: Superiority; estimated/derived from the number of dos = 30 — This trial had a 3+3 study design. Escalation/de-escalation through cohorts were based on DLT events. MTD based on DLT events was determined to be 30mg; 30 mg

2. Secondary Outcome: Count of Participants Who Did Not Experience a DLT Are Listed in the Outcome Measure Data Table
Description: A RP2D equal to or less than the MTD will be declared after the MTD is determined and will be used for the Dose Expansion Phase, if conducted. After the RP2D is determined, a dose expansion phase, of up to 10 additional patients, might be conducted, in which a preliminary determination of efficacy will be conducted, using the ELN criteria.
Time Frame: 28 days
Population: No descalation cohort less than cohort 1 dose was needed. Due to DLTs, no patients enrolled to cohort 4 or 5.
Measure: Count of Participants; unit: Participants
Arm/Group | De-escalation Cohort; 20mg | Cohort 1; 30 mg | Cohort 2; 40mg | Cohort 3; 60mg | Cohort 4; 80mg | Cohort 5; 100mg
Number analyzed (Participants) | 0 | 5 | 7 | 4 | 0 | 0
Participants | 0 | 5 | 5 | 2 | 0 | 0
Statistical Analysis 1: Comparison: De-escalation Cohort; 20mg vs Cohort 1; 30 mg vs Cohort 2; 40mg vs Cohort 3; 60mg vs Cohort 4; 80mg vs Cohort 5; 100mg; Test type: Superiority; estimated/derived from the number of = 30 — This trial had a 3+3 study design. Escalation/de-escalation through cohorts were based on DLT events. Established recommended phase 2 dose (RP2D) was determined to be 30mg; 30 mg

ADVERSE EVENTS:
Time Frame: Adverse Events will be reported and recorded in the eCRF from the time of the first dose of study drug through 30 days after the last dose of study drug or until the start of subsequent antineoplastic therapy, whichever occurs first. This is patient-dependent based on the # of cycles they complete, with an average of 1 cycle completed or approximately 58 days to report Adverse Events.
Description: 1. All-Cause Mortality
  2. Serious Adverse Events
  3. Other (Not Including Serious) Adverse Events
Arm/Group | De-escalation Cohort; 20mg | Cohort 1; 30 mg | Cohort 2; 40mg | Cohort 3; 60mg | Cohort 4; 80mg | Cohort 5; 100mg
All-Cause Mortality (participants affected / at risk) | 0/0 | 5/5 | 6/7 | 4/4 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 2/5 | 3/7 | 3/4 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 5/5 | 7/7 | 4/4 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | De-escalation Cohort; 20mg (N=0) | Cohort 1; 30 mg (N=5) | Cohort 2; 40mg (N=7) | Cohort 3; 60mg (N=4) | Cohort 4; 80mg (N=0) | Cohort 5; 100mg (N=0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Covid-19 Infection
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — C. diff infection
Lung infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | De-escalation Cohort; 20mg (N=0) | Cohort 1; 30 mg (N=5) | Cohort 2; 40mg (N=7) | Cohort 3; 60mg (N=4) | Cohort 4; 80mg (N=0) | Cohort 5; 100mg (N=0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (16) | 4 (16) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 4 (5) | 3 (4) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Haptoglobin Increase
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Protein Total Serum Decreased
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Uric Acid Decreased
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — White Blood Cell Increased
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA — Chloride Serum Increased
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — Monocytes Decreased
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — Increased Cardiac Troponin I
Blood bicarbonate decreased (Investigations) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA
Blood bilirubin increased (Investigations) | NA | 2 (4) | 0 (0) | 1 (1) | NA | NA
Blood lactate dehydrogenase increased (Investigations) | NA | 2 (3) | 0 (0) | 0 (0) | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA
Bruising (Injury, poisoning and procedural complications) | NA | 0 (0) | 1 (1) | 1 (1) | NA | NA
Cardiac arrest (Cardiac disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Cardiac disorders - Other, specify (Cardiac disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — CPK Decrease
Constipation (Gastrointestinal disorders) | NA | 2 (2) | 2 (2) | 0 (0) | NA | NA
Cough (General disorders) | NA | 1 (2) | 0 (0) | 1 (1) | NA | NA
Cystitis noninfective (Renal and urinary disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Depression (Psychiatric disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Device related infection (Infections and infestations) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Diarrhea (Gastrointestinal disorders) | NA | 1 (1) | 3 (3) | 1 (1) | NA | NA
Dizziness (Immune system disorders) | NA | 1 (1) | 2 (2) | 0 (0) | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | NA | 1 (2) | 0 (0) | 0 (0) | NA | NA
Eczema (Skin and subcutaneous tissue disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Edema limbs (General disorders) | NA | 1 (1) | 3 (3) | 3 (5) | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA
Erythema multiforme (Skin and subcutaneous tissue disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Eye disorders - Other, specify (Eye disorders) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA — scleral icterus
Eye disorders - Other, specify (Eye disorders) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA — Posterior Vitreus Detachment
Fall (Injury, poisoning and procedural complications) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Fatigue (General disorders) | NA | 4 (5) | 3 (3) | 1 (1) | NA | NA
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA — blackening gums
General disorders and administration site conditions - Other, specify (General disorders) | NA | 1 (1) | 2 (2) | 0 (0) | NA | NA — Appetite change
General disorders and administration site conditions - Other, specify (General disorders) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA — mild nasal swelling
General disorders and administration site conditions - Other, specify (General disorders) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA — toenail fungus
General disorders and administration site conditions - Other, specify (General disorders) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA — carbon dioxide decrease
General disorders and administration site conditions - Other, specify (General disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — bleeding gums
General disorders and administration site conditions - Other, specify (General disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — activity change
General disorders and administration site conditions - Other, specify (General disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — forgetfulness
General disorders and administration site conditions - Other, specify (General disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — Intermittent decreased total protein
General disorders and administration site conditions - Other, specify (General disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — left leg edeuma
General disorders and administration site conditions - Other, specify (General disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — lightheadedness
General disorders and administration site conditions - Other, specify (General disorders) | NA | 0 (0) | 1 (2) | 0 (0) | NA | NA — Arthralgia
General disorders and administration site conditions - Other, specify (General disorders) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA — decreased protein
General disorders and administration site conditions - Other, specify (General disorders) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA — increased chlorine
Generalized edema (General disorders) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA
Hallucinations (Psychiatric disorders) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA
Hyperglycemia (Metabolism and nutrition disorders) | NA | 0 (0) | 2 (3) | 1 (1) | NA | NA
Hyperkalemia (Metabolism and nutrition disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Hypermagnesemia (Metabolism and nutrition disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Hyperphosphatemia (Metabolism and nutrition disorders) | NA | 0 (0) | 2 (2) | 0 (0) | NA | NA
Hyperuricemia (Metabolism and nutrition disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | NA | 1 (1) | 1 (1) | 0 (0) | NA | NA
Hypocalcemia (Metabolism and nutrition disorders) | NA | 1 (3) | 5 (5) | 3 (4) | NA | NA
Hypoglycemia (Metabolism and nutrition disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | NA | 0 (0) | 3 (3) | 1 (3) | NA | NA
Hypomagnesemia (Metabolism and nutrition disorders) | NA | 0 (0) | 2 (2) | 0 (0) | NA | NA
Hyponatremia (Metabolism and nutrition disorders) | NA | 2 (3) | 2 (3) | 0 (0) | NA | NA
Hypophosphatemia (Metabolism and nutrition disorders) | NA | 0 (0) | 0 (0) | 2 (2) | NA | NA
Hypotension (Vascular disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA
Ileus (Gastrointestinal disorders) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA
Investigations - Other, specify (Investigations) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA — BUN Increased
Investigations - Other, specify (Investigations) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA — activity change
Investigations - Other, specify (Investigations) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA — Appetite change (Poor appetite)
Investigations - Other, specify (Investigations) | NA | 1 (3) | 0 (0) | 0 (0) | NA | NA — aspartate aminotransferase decrease
Investigations - Other, specify (Investigations) | NA | 1 (1) | 1 (1) | 0 (0) | NA | NA — hyperbilirubinemia
Investigations - Other, specify (Infections and infestations) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA — joint swelling
Investigations - Other, specify (Investigations) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA — mouth sores
Investigations - Other, specify (Investigations) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — pneumonia
Investigations - Other, specify (Investigations) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — post arrest mixed shock
Investigations - Other, specify (Investigations) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — subarachinoid hemorrhage
Lung infection (Infections and infestations) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA — Creatinine Decrease (Intermittent)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA — increased chloride
Myalgia (Musculoskeletal and connective tissue disorders) | NA | 3 (5) | 2 (2) | 0 (0) | NA | NA
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA — Right Sided Hip Pain
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — Bilateral Wrist Edema
Nausea (Gastrointestinal disorders) | NA | 1 (1) | 0 (0) | 1 (1) | NA | NA
Nervous system disorders - Other, specify (Nervous system disorders) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA — lightheadedness
Neutrophil count decreased (Investigations) | NA | 2 (12) | 3 (6) | 0 (0) | NA | NA
Oral hemorrhage (Gastrointestinal disorders) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Platelet Count Decrease (Investigations) | NA | 4 (34) | 5 (13) | 0 (0) | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1) | 1 (1) | 0 (0) | NA | NA
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | NA | 1 (1) | 1 (1) | 1 (1) | NA | NA
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA — Intermittent Tachypnea
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA — interstitial lung disease
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — acute respiratory failure
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — right sided pleural effusion
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA — Covid-19 Infection
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA — Epistaxis
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA — Rales
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1) | 1 (1) | 0 (0) | NA | NA
Sepsis (Infections and infestations) | NA | 1 (1) | 2 (2) | 1 (1) | NA | NA
Sinus tachycardia (Cardiac disorders) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA — 0.5 cm nodule (right anterior thigh)
Skin infection (Infections and infestations) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Sore throat (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA
Stomach pain (Gastrointestinal disorders) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA
Thromboembolic event (Vascular disorders) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Thrush (Infections and infestations) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA
Thyroid stimulating hormone increased (Investigations) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Tooth infection (Infections and infestations) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA
Urinary tract infection (Infections and infestations) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Urine output decreased (Investigations) | NA | 0 (0) | 1 (1) | 0 (0) | NA | NA
Vomiting (Gastrointestinal disorders) | NA | 0 (0) | 0 (0) | 1 (1) | NA | NA
Weight loss (Investigations) | NA | 1 (1) | 0 (0) | 0 (0) | NA | NA
White blood cell decreased (Investigations) | NA | 1 (5) | 3 (6) | 0 (0) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-29): https://cdn.clinicaltrials.gov/large-docs/45/NCT04914845/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT04914845/ICF_001.pdf